CLINICAL TRIAL: NCT01767792
Title: Open-label, Phase 2 Study of Bevacizumab in Children and Young Adults With Neurofibromatosis 2 and Progressive Vestibular Schwannomas That Are Poor Candidates for Standard Treatment With Surgery or Radiation
Brief Title: Phase 2 Study of Bevacizumab in Children and Young Adults With NF 2 and Progressive Vestibular Schwannomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF4807; W81XWH-12-1-0155 (Other Grant/Funding Number: Dept. of Defense - US Army)
Record Dates: First submitted 2013-01-07; First posted 2013-01-14 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Neurofibromatosis Type 2; Progressive Vestibular Schwannomas
Keywords: Neurofibromatosis Type 2; Progressive Vestibular Schwannomas
MeSH Terms: conditions — Neurofibromatosis 2 | interventions — Bevacizumab; Vascular Endothelial Growth Factor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Follow participant for 2 years and assess hearing response rates
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Treatment will be administered on an outpatient basis. Bevacizumab is administered by IV infusion at a dose of 10 mg/kg every 2 weeks for 24 weeks (induction therapy, see Schema). One cycle lasts 28 days and includes two infusions of bevacizumab. Clinical response will be assessed by audiology and MRI at weeks 12 and 24. Subjects with hearing decline at weeks 12 and 24 will be taken off of protocol. After week 24, patients with a clinical response or stable disease (together comprising "clinical benefit") will transition to maintenance therapy with bevacizumab.
  During the maintenance phase, subjects will be treated with open-label bevacizumab 5 mg/kg every 3 weeks for up to 72 weeks. Subjects will be followed with audiology and MRI scans every 12 weeks. The total time of the study will be 96 weeks (24 weeks induction + 72 weeks maintenance).
  Other Names: rhuMAb; Vascular Endothelial Growth Factor (VEGF); Avastin®

SUMMARY:
To determine the hearing response rate at 24 weeks after treatment with bevacizumab for symptomatic vestibular schwannomas (VS) in children and young adults with Neurofibromatosis Type 2 (NF 2).

DETAILED DESCRIPTION:
Subjects will be treated with open-label bevacizumab 10 mg/kg every 2 weeks for 24 weeks (induction therapy). Clinical response will be assessed by audiology and MRI at weeks 12 and 24. Subjects with hearing decline at weeks 12 or 24 will be taken off of protocol. At week 24, patients with a clinical response or stable disease (together comprising "clinical benefit") will transition to maintenance therapy with bevacizumab. During the maintenance phase, subjects will be treated with open-label bevacizumab 5 mg/kg every 3 weeks for up to 72 weeks. Subjects will be followed with audiology and MRI scans every 12 weeks. The total time of the study will be 96 weeks (24 weeks induction + 72 weeks maintenance).

Subjects will be allowed to increase their bevacizumab dose to 10 mg/kg every 2 weeks during maintenance therapy if they experience hearing decline during maintenance therapy (defined as decrease in word recognition score below the 95% critical difference compared with the word recognition score at baseline, Appendix A). Subjects will be taken off of study if their word recognition score does not remain within the 95% critical difference after receiving bevacizumab 10 mg/kg every 2 weeks.

ELIGIBILITY:
Inclusion Criteria - Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Patients must have a confirmed diagnosis of neurofibromatosis 2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria, or by detection of a causative mutation in the Neurofibromatosis 2 (NF2) gene.
* Patients must have measurable disease, defined as at least one VS > 1.0 ml (on volumetric analysis) that can be accurately measured by contrast-enhanced cranial MRI scan with fine cuts through the internal auditory canal (3 mm slices, no skip).
* Age 6 years or greater (no upper limit) on day 1 of treatment. Given the potential risk of long-term bevacizumab use, children under age 6 are not eligible for treatment. No upper limit for adults.
* Life expectancy of greater than 1 year.
* Karnofsky performance status ≥ 70.
* Participants must have normal organ and marrow function as defined below with definitions micro liter (mcL), Aspartate aminotransferase (AST), Serum glutamic oxaloacetic transaminase (SGOT), Alanine aminotransferase (ALT), Serum glutamic pyruvic transaminase (SGPT):
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
* Patients must have a creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥60ml/min/1.73 m2 or a normal serum creatinine based on age described in the table below:
* Age Maximum Serum Creatinine (mg/dL) 6 to < 10 years 1(Male) 1(Female) 10 to < 13 years 1.2(Male) 1.2(Female) 13 to < 16 years 1.5(Male) 1.4(Female

  ≥ 16 years 1.7(Male) 1.4(Female)
* Subjects must have a target VS with the following qualities:
* Not amenable to surgery due to patient refusal, high risk for surgical complications (e.g., damage to lower cranial nerve function, tumor size > 3 cm in longest diameter, or multilobulated tumor appearance on MRI scan).
* Associated with a word recognition score of < 85%
* Documented clinical progression defined as EITHER:
* Progressive hearing loss (defined as a decline in word recognition score below the 95% critical difference interval from baseline score [Appendix A] related to VS (i.e., not due to prior interventions such as surgery or radiation)

OR

* Progressive tumor growth in the preceding 18 months, defined as ≥ 20% increase in volume
* The effects of bevacizumab on the developing human fetus are unknown. For this reason and because bevacizumab agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign written informed consent and assent documents.
* Must have established relationship with primary care physician and provide contact information

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Prior radiation treatment to the target vestibular schwannoma is allowed if provided 3 years prior to participation in the clinical trial. Prior radiation treatment to non-target tumors is allowed.
* Participants may not be receiving any other study agents.
* Patients with nervous system tumors associated with NF2 (e.g., schwannomas, meningiomas, ependymomas, or gliomas) will not be excluded from this clinical trial unless (in the opinion of the investigator) these tumors are growing and are likely to require treatment during the clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab.
* Patients with known hypersensitivity of Chinese hamster ovary cell products, other recombinant human antibodies, or compounds of similar chemical or biologic composition to bevacizumab.
* Inability to tolerate periodic MRI scans or gadolinium contrast.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of arterial/myocardial disease.
* Clinically significant cardiovascular disease, such as:
* Inadequately controlled hypertension (HTN) (for adults: Systolic Blood Pressure (SBP) > 160 mmHg and/or Diastolic Blood Pressure (DBP) > 90 mmHg despite antihypertensive medication; for children: please refer to Appendix D for age-appropriate values indicating ≥ Grade 2)
* History of cerebrovascular accident (CVA) within 12 months
* Myocardial infarction or unstable angina within 12 months
* New York heart association grade II or greater congestive heart failure
* Serious and inadequately controlled cardiac arrhythmia
* Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection)
* Clinically significant peripheral vascular disease
* Pregnant women are excluded from this study because bevacizumab is an anti-angiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with bevacizumab, breastfeeding should be discontinued if the mother is treated with bevacizumab. These potential risks may also apply to other agents used in this study.
* HIV-positive patients or cancer survivors are eligible for this study if they fulfill all other eligibility criteria.
* Concurrent use of anti-coagulant drugs (not including prophylactic doses), history of coagulopathy, or evidence of bleeding diathesis or coagulopathy.
* Imaging (CT or MRI) evidence of hemorrhage deemed significant by the treating physician (> grade 1). Subjects with history of central nervous system (CNS) hemorrhage are not eligible.
* Urine protein should be screened by urine analysis for Urine Protein Creatinine (UPC) ratio. For UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be <1000 mg for patient enrollment.
* Serious or non-healing wound, ulcer or bone fracture.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1.
* Invasive procedures defined as follows:
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
* Brain biopsy within 28 days prior to day 1 of therapy (wounds must be fully healed from brain biopsies performed more than 28 days prior to day 1 of therapy)
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to D1 therapy
* Prior treatment with bevacizumab.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plotkin, MD, Study Chair — Massachusetts General Hospital
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's HealthCare of Atlanta, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana Unversity, Indianapolis, Indiana
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Children' Hospital Boston and Massachusetts General Hospital, Boston, Massachusetts
  - Washington University - St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Safety and tolerability of bevacizumab for 2 years. Change in hearing response will also be monitored.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab: Follow participant for 2 years and assess hearing response rates
  Bevacizumab: Treatment will be administered on an outpatient basis. Bevacizumab is administered by IV infusion at a dose of 10 mg/kg every 2 weeks for 24 weeks (induction therapy, see Schema). One cycle lasts 28 days and includes two infusions of bevacizumab. Clinical response will be assessed by audiology and MRI at weeks 12 and 24. Subjects with hearing decline at weeks 12 and 24 will be taken off of protocol. After week 24, patients with a clinical response or stable disease (together comprising "clinical benefit") will transition to maintenance therapy with bevacizumab.
  During the maintenance phase, subjects will be treated with open-label bevacizumab 5 mg/kg every 3 weeks for up to 72 weeks. Subjects will be followed with audiology and MRI scans every 12 weeks. The total time of the study will be 96 weeks (24 weeks induction + 72 weeks maintenance).
Arm/Group | Bevacizumab
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Participants enrolled in the United States
  participants
    United States | 22
Word recognition score in target ear [Median (Full Range); unit: number correct words] | 53 [6 to 82]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Hearing
Description: Number of participants with a statistically significant increase in word recognition score on audiology compared to baseline.
Time Frame: 6 months
Population: All participants treated with bevacizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab: Induction (high dose) therapy.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 22
Participants | 9

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events occurring in at least 10% of participants during induction therapy.
Time Frame: 6 months
Population: All participants treated with bevacizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 22
Participants | 22

3. Secondary Outcome: Tolerability of Bevacizumab During Induction (High Dose) Therapy
Description: Number of participants who did not stop treatment due to side effects or by participant/provider choice during induction period.
Time Frame: 6 months
Population: All participants treated with bevacizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 22
Participants | 21

4. Secondary Outcome: Durability of Hearing Response During Maintenance (Low Dose) Therapy
Description: Number of participants with hearing improvement during induction therapy who maintained hearing improvement relative to baseline during maintenance therapy as measured by word recognition score.
Time Frame: 2 years
Population: Analysis population is restricted to participants who achieved hearing improvement during induction (high dose) therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab: Maintenance (low dose) therapy.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 7
Participants | 4

5. Secondary Outcome: Changes in Pure Tone Average (PTA) on Audiology Compared With Baseline, Measured in Decibels (dBHL).
Description: Increase in pure tone average represents worsening of hearing and decrease in pure tone average represents improvement of hearing. Range for for pure tone average (PTA) is 0-110 dBHL (decibels).
Time Frame: Weeks 25, 49, 73, 98
Population: All participants treated during maintenance (low dose) therapy.
Measure: Least Squares Mean (Standard Error); unit: decibels (dBHL)
Arm/Group | Bevacizumab
Number analyzed (Participants) | 20
decibels (dBHL)
  Change from week 25 to week 49 | -1.19 (1.91)
  Change from week 25 to week 73 | 1.05 (1.91)
  Change from week 25 to week 98 | -0.95 (2.09)

6. Secondary Outcome: Changes in Distress Related to Tinnitus During Induction (High Dose) Treatment.
Description: Self-reported distress measured using the tinnitus reaction questionnaire (TRQ). TRQ has 26 questions measured on a 5-point Likert scale from 0 (not at all) to 4 (almost all of the time). The total score is the sum of the responses with higher scores indicating more reported distress.
Time Frame: 6 months (induction phase)
Population: Number of participants with data at baseline and month 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab
Number analyzed (Participants) | 21
units on a scale | 14.3 (18.2)

7. Secondary Outcome: Durability of Radiographic Response
Description: Count of participants who achieved a 20% or more reduction in tumor volume over baseline during induction (high dose) therapy and maintained this decrease during maintenance (low dose) therapy (decline in tumor volume from baseline of 20% or more).
Time Frame: 2 years
Population: Analysis population is restricted to participants who achieved hearing improvement during induction (high dose) therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 7
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse event data collected for 2 years
Arm/Group | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=22)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=22)
Hypertension (Vascular disorders) | 11 (28)
Fatigue (Nervous system disorders) | 8 (17)
Headache (Nervous system disorders) | 7 (13)
Irregular menstruation (Reproductive system and breast disorders) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 4 (5)
Proteinuria (Renal and urinary disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
AST increased (Investigations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT01767792/Prot_SAP_ICF_000.pdf